CLINICAL TRIAL: NCT02990052
Title: Conservative Treatment vs. Volar Plating of Distal Radius Fractures in Patients Aged Over 50 Years Old: A Prospective Randomized Trial
Brief Title: Conservative Treatment vs. Volar Plating of Distal Radius Fractures
Acronym: DRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Distal Radius Fr. Sirniö
Record Dates: First submitted 2016-11-07; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volar plating (Active Comparator): Volar fixed-angle plating for dislocated distal radius fracture after closed reduction.
  Interventions: Procedure: Volar plating
- Conservative treatment (Active Comparator): Primary conservative treatment (closed reduction and casting) for dislocated distal radius fracture.
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Volar plating — Open reduction and volar fixed-angle plate fixation of distal radius fracture
  Arms: Volar plating
Procedure: Conservative treatment — Closed reduction & casting of distal radius fracture
  Arms: Conservative treatment

SUMMARY:
A prospective, randomized controlled single-center trial with 80 patients aged 50 years and above to compare the functional and radiological results of conservative treatment and volar fixed-angle plating in the management of distal radius fracture

DETAILED DESCRIPTION:
Volar plating has became as a standard approach for treating unstable distal radius fractures. The incidence of surgically treated patients with distal radius fractures has increased many fold from the beginning of this millennium, owing mostly to increased number of volar platings. The most striking increase of plate fixations has occurred in older patient groups, especially in females. With volar fixed-angle plate, very near-anatomic, stable fixation with relatively low complication rate, can be achieved even in osteoporotic bone. There are only few randomized, prospective studies comparing results of volar plating and conservative treatment, comparing patients aged over 65 years. Quite little is known of the results comparing conservative treatment and volar plating in patients aged below 65 years.

Main goal of our study was to compare the functional and radiological results of conservative treatment and volar fixed-angle plating in the management of distal radius fracture in patients aged over 50 years an older.

ELIGIBILITY:
Inclusion Criteria:

* patients over 50 years-old
* primary dislocated distal radius fracture (AO/OTA 23 type A2-3 and C1-2)
* primary reduction of fracture is acceptable considering primary conservative treatment

Exclusion Criteria:

* bilateral and open fractures and fractures with neurovascular compromise
* other major concurrent fracture necessitating treatment of any kind
* patients under 50 years of age
* previous ipsilateral distal radius fracture
* inflammatory joint disease
* significant radiocarpal-joint degeneration
* patient's bad co-operation or major co-morbidity making an operation contraindicated

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-11; Primary Completion 2014-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Difference of DASH-score between two study groups | 2 year observation
  Disability of the Arm, Shoulder and Hand -Score assessing the function of the upper extremity

SECONDARY OUTCOMES:
Difference of radiological parameters between two study groups | 2 year observation
  Dorsal angulation, ulnar variance and radial inclination of distal radius. Osteoarthritis of radiocarpal joint

IPD SHARING:
Plan to Share IPD: Undecided